CLINICAL TRIAL: NCT02536781
Title: Khon Kaen University Ethics Committee in Human Research
Brief Title: Efficacy of Anthocyanin Mouthrinse for Oral Anti-inflammation From Orthodontic Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sucharat Limsitthichaikoon, Pharmaceutical Technology, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE582088
Record Dates: First submitted 2015-08-22; First posted 2015-09-01 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Inflammation of Mouth; Acute Mucous Inflammation
Keywords: Anthocyanin; Inflammation; Orthodontic treatment
MeSH Terms: conditions — Stomatitis; Inflammation | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebol (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Anthocynin (Active Comparator): Anthocyanin
  Interventions: Drug: Anthocyanin

INTERVENTIONS:
Drug: Anthocyanin — Anti-inflammation gel
  Arms: Anthocynin
Drug: Placebo — Blank gel
  Arms: Placebol

SUMMARY:
The purpose of this study is to compare the oral inflammatory reduction effect caused from orthodontic treatment of anthocyanin and placebo mouthrinse.

DETAILED DESCRIPTION:
Multiple inflammatory lesions caused from orthodontic treatments are commonly found in these patients and the irritations from the insertion of the orthodontic wire are hard to apply the topical cream or gel. Standard treatment to prevent oral mucosal irritation caused from orthodontic brackets and wires is an orthodontic wax to cover the appliances. However, the covering wax is just a prophylactic measure to protect the mucosal irritation. Thus, the patients still need a specific treatment for their oral inflammatory condition. Developing a product that can treat entire inflammatory areas in oral cavity, promote oral hygiene, and anti-fungal would be beneficial and useful for the orthodontic treatment. Anthocyanins, one of a natural compound from red, blue, purple vegetables, fruits, and flowers, have many beneficial effects including anti-inflammation and the most important effect superior to steroid usage is anti-candidiasis. Interesting in anthocyanins as the natural treatment, has drawn attention due to the benefits in oral inflammation. Previous study on the effect of a topical anthocyanin gel demonstrated positive effect of topical anthocyanins gel against oral inflammation in human subjects at 6 weeks. Unfortunately, anthocyanin is not stable and easily to be degraded. Therefore, stabilized anthocyanin oral formulation needs to be developed and the formulation needs to provide stable and active anthocyanins in suitable oral formula. This study aims to prepare and investigate effects of anthocyanin complex in order to formulate the mouthrinse for anti-inflammation caused by orthodontic treatment. Thus, to prepare and investigate the effects of anthocyanin activities after forming complexation in order to formulate the mouthrinse would be evaluated. In addition, the examination of anti-oral inflammation caused by orthodontic treatment by anthocyanin complex in clinical trial will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or females between the ages of 18 and 35 with oral inflammation, investigated by a dentist, caused by orthodontic devices.
* The inflammatory lesions are occurred at labial and/or buccal mucosa.
* Be able to communicate well with the investigator and to comply with the requirements of the entire study.
* Not participate in other project(s).
* Be willingness to give written informed consent (prior to any study-related procedures being performed) and to be able to adhere to the study restrictions and examination schedule.

Exclusion Criteria:

* - Have the persistent inflammatory lesions and/or ulcers that cannot be healed more than 2 weeks or the inflammation that may lead to be oral cancer.
* Have severe oral inflammation or the inflammation occur from ongoing head and neck chemotherapy or serious oral inflammatory such as periodontitis and oral lichen planus.
* Taking steroid or applying topical steroid within or 7 days before participated in this study.
* Have a history of allergy or hypersensitivity to any red, blue, or purple color fruits and vegetables such as berry groups.
* Patients with auto-immune diseases or diseases that related to wound healing process such as diabetes.
* Patients that cannot meet the follow up or drop out of the experiments.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sucharat Limsitthichaikoon, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Maung, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Nizamutdinova IT, Kim YM, Chung JI, Shin SC, Jeong YK, Seo HG, Lee JH, Chang KC, Kim HJ. Anthocyanins from black soybean seed coats stimulate wound healing in fibroblasts and keratinocytes and prevent inflammation in endothelial cells. Food Chem Toxicol. 2009 Nov;47(11):2806-12. doi: 10.1016/j.fct.2009.08.016. Epub 2009 Sep 4. PMID 19733615
- [Result] Shumway BS, Kresty LA, Larsen PE, Zwick JC, Lu B, Fields HW, Mumper RJ, Stoner GD, Mallery SR. Effects of a topically applied bioadhesive berry gel on loss of heterozygosity indices in premalignant oral lesions. Clin Cancer Res. 2008 Apr 15;14(8):2421-30. doi: 10.1158/1078-0432.CCR-07-4096. PMID 18413833

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Mucoadhesive gel without any drug or treatment. Apply 2 time daily (Morning and Night)
- Anthocynin: Mucoadhesive gel containing 10% of anthocyanin complex. Apply 2 times daily (Morning and night)
Period: Overall Study
Arm/Group | Placebo | Anthocynin
Started | 36 | 34
Completed | 34 | 34
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebol: Blank gel
  Anthocyanin: Anti-inflammation gel
- Anthocynin: Anthocyanin gel
  Placebo: Blank gel
- Total: Total of all reporting groups
Arm/Group | Placebol | Anthocynin | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (1.5) | 22.4 (1.6) | 22.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  Thailand | 36 | 34 | 70
VAS scores range from 0 (no pain) to 10 (severe pain) [Mean (Standard Deviation); unit: scores on a scale] | 3.6 (1.8) | 3.6 (1.7) | 3.6 (1.7)
wound area [Mean (Standard Deviation); unit: mm^2] | 33.3 (37.8) | 26.5 (32.2) | 29.08 (35.01)

OUTCOME MEASURES:

1. Primary Outcome: Wound Size (mm^2) Reduction
Description: Comparing between the active and placebo about the wound size reduction from day 0 to day 7 after treatment
Time Frame: Days 0 and 7 after treatment
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Placebol | Anthocynin
Number analyzed (Participants) | 34 | 34
mm^2 | 11.26 (14.22) | 8.92 (14.86)

2. Secondary Outcome: VAS Scores Range From 0 (no Pain) to 10 (Severe Pain)
Time Frame: Days 0 and 7 after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebol | Anthocynin
Number analyzed (Participants) | 34 | 34
units on a scale | 1.53 (1.67) | 0.96 (0.68)

ADVERSE EVENTS:
Time Frame: The participants were monitored adverse event for 8 days (in the periods of the experiments (7 days) and followed up after the last visit for 24 hour, which total observation of the adverse event equal 8 days)
Description: "70 participants may be in risks, but all participants, that we monitored, found no adverse events
Groups:
- Placebol: Placebo gel
  Placebo gel
- Anthocynin: Anthocyanin gel
  Anti-inflammation gel
Arm/Group | Placebol | Anthocynin
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No